CLINICAL TRIAL: NCT04573907
Title: Comparative Bioavailability Study of Levothyroxine Sodium Tablets 100 mcg in Healthy Volunteers
Brief Title: Bioequivalence Study of Levothyroxine Sodium Tablets 100 mcg
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tecnoquimicas (Industry)
Collaborators: DominguezLab (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PRO-BEQ-LEVO-007-V.01
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Formulation of Levothyroxine (Experimental): Levothyroxine sodium tablets 100 mcg Single dose of 600 mcg administered in dosing period 1 or 2
  Interventions: Drug: Drug Levothyroxine 100 mcg
- Reference formulation of Levothyroxine (Active Comparator): Eutirox 100 mcg Single dose of 600 mcg administered in dosing period 1 or 2
  Interventions: Drug: Drug Eutirox 100 mcg

INTERVENTIONS:
Drug: Drug Levothyroxine 100 mcg — Administration of a 600 mcg levothyroxine dose
  Arms: Test Formulation of Levothyroxine
Drug: Drug Eutirox 100 mcg — Administration of a 600 mcg levothyroxine dose
  Arms: Reference formulation of Levothyroxine

SUMMARY:
The objective of this study is to establish the bioequivalence of two levothyroxine formulations through the estimation of T4 levels in serum samples after baseline correction, according to Food and Drugs Administration (FDA), World Health Organization (WHO) and Colombian National Vigilance Institute for Drugs and Food (INVIMA) guidelines.

DETAILED DESCRIPTION:
Levothyroxine (T4) is used to treat patients with hypothyroidism and may often result in lifelong therapy. Its physiologically active metabolite is tri-iodothyronine (T3). Levothyroxine is also endogenously produced in the body. Since small changes in levothyroxine administration (e.g. change in brand or formulation) can cause significant changes in serum thyroid stimulating hormone (TSH) concentrations, precise and accurate TSH control is critical to avoid potential adverse iatrogenic effects. Tecnoquimicas modified its Levothyroxine tablets formulation in order to comply with new pharmacopeial specifications. It will then evaluate the impact on drug product performance based on pharmacokinetic (PK) measures of total serum T4 and total serum T3 of the new formulation of levothyroxine (Test formulation) relative to the reference formulation from Merck (Reference formulation)

This will be a single-center, open-label, two-period, two-treatment, two-sequence, randomized, single-dose, crossover study. 80 healthy adults will be randomized to receive a single dose (6 x 100 mcg tablets = 600 mcg) of the test formulation of levothyroxine and reference formulation of levothyroxine separately in each treatment period. There will be two treatment sequences (AB, BA) and a 42 day washout between the two treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Healthy volunteers according to antecedents, clinical evaluation, biochemical tests and other complimentary tests
* Sex: both (male and female, homogenously distributed)
* Age: 18 to 50 years old
* BMI: 18 to 30 kg/m2
* Non smokers from at least 3 months

Exclusion Criteria:

* History of liver disease, kidney disease or conditions of psychiatric origin.
* History of drug or alcohol abuse in the last two years.
* Ingestion of other drugs the 2 weeks prior to the start of the study.
* History of seizure disorders, depressive disorders, cardiovascular diseases, hematological, metabolic, vesicular or other, that the Principal Investigator judges clinically significant.
* Abnormal electrocardiogram (EKG).
* Hypersensitivity to Levothyroxine sodium or to excipients (from formulations to test).
* Positive HIV test; hepatitis B and C.
* Positive urine drug dose of abuse.
* Having participated in another research study in the last 6 months.
* Having donated blood within the 3 months prior to the start of the study.
* Clinically significant abnormal laboratory test results.
* Abnormal results outside the reference values for thyroid function (T3, T4, TSH, anti-TPO antibodies).
* Female volunteers who are breastfeeding during the study period.
* Positive beta-HCG test in female volunteers.
* Volunteers who must start a scheduled medical or pharmacological treatment outside the this Protocol.
* Volunteers who do not maintain the conditions of fasting and food intake in the pre-established schedules.
* Volunteers who do not avoid the intake of coffee, tea, grapefruit, cola and / or alcoholic beverages during the 48 h preceding the study.
* Volunteers on a special diet in the last 28 days (eg vegetarian diet, etc.).
* Volunteers with clinically significant allergies to food, medication, etc.
* Non-cooperative volunteers.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
(AUC) Area Under the Curve 0-48 for T4 | [Time Frame: From 0 to 48 hours]
  -30 min., -15 min., 0 hour (h ) pre-dose; 30 min., 1 h, 1.30 h, 2 h, 2.30 h, 3 h, 4 h, 6 h, 8 h, 10 h, 12 h, 16 h, 24 h , 48 hours
(Cmax) Maximum concentration 0-48 for T4 | [Time Frame: From 0 to 48 hours]
  -30 min., -15 min., 0 hour ( h) pre-dose; 30 min., 1 h, 1.30 h, 2 h, 2.30 h, 3 h, 4 h, 6 h, 8 h, 10 h, 12 h, 16 h, 24 h , 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- DominguezLab, Paraná, Entre Ríos Province, Argentina

IPD SHARING:
Plan to Share IPD: No